CLINICAL TRIAL: NCT02710643
Title: "MIRO" (Molecularly Oriented Immuno - Radio -Therapy): Multicenter Phase II Study for the Treatment of the Molecular Basis of Stage I / II Follicular Lymphoma With Local Radiotherapy With / Without Ofatumumab
Brief Title: "MIRO" Molecularly Oriented Immuno-radio-therapy
Acronym: FIL_MIRO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIL_MIRO
Record Dates: First submitted 2016-02-26; First posted 2016-03-17 (Estimated); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Follicular Lymphoma, Grade 1; Follicular Lymphoma, Grade 2; Follicular Lymphoma Grade 3A
Keywords: Follicular; Lymphoma; Grade 1; Grade 2; Grade 3A
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma | interventions — ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- MRD - BEFORE RT (No Intervention): Patients who had negative baseline Bcl-2 in PB and BM will not undergo further treatment after radiotherapy; they will not repeat Bcl-2 during subsequent follow-up visits.
- MRD + BEFORE RT AND MRD - AFTER RT (No Intervention): Patients who had positive baseline Bcl-2 in PB and / or BM and become negative after local radiotherapy will not undergo further treatment.
- MRD + BEFORE RT AND MRD + AFTER RT (Experimental): Patients who had positive baseline Bcl-2 in PB and / or BM and remain positive after local radiotherapy get Ofatumumab (8 weekly infusion of 1000 mg total dose).
  Patients Bcl-2 negativized either after radiotherapy or after Ofatumumab, who became Bcl-2 positive during the follow-up monitoring will be treated/retreated with Ofatumumab 8 weekly infusions at the conventional dose of 1000 mg; Bcl-2 monitoring will be continued subsequently according to the program.In case of persistent positive PCR after Ofatumumab the treatment will not be repeated.
  Interventions: Drug: OFATUMUMAB

INTERVENTIONS:
Drug: OFATUMUMAB — 8 weekly infusion of 1000 mg total dose
  Other Names: ARZERRA
  Arms: MRD + BEFORE RT AND MRD + AFTER RT

SUMMARY:
Phase II prospective multicenter study for stage I/II Follicular Lymphoma treated with involved-field radiotherapy (IFRT) at doses of 24 Gy) with or without Ofatumumab for 8 weekly doses on molecular basis. Patients with positive basal Bcl-2 will be followed every 3 months and with Bcl-2 detection every 6 months for 3 years. Patient with negative basal Bcl-2 will be followed every 3 months without further Bcl-2 detection.

Ofatumumab treatment will be administered to:

1. Patients with positive basal PCR for Bcl-2-IgH rearrangement in BM and/or PB, resulting still positive after IFRT;
2. Patients with positive basal PCR for Bcl-2-IgH in

DETAILED DESCRIPTION:
Stage I/IIA follicular lymphoma (FL) is considered a localized disease that can be adequately treated with radiotherapy alone. This strategy is recommended by the guidelines of the "Società Italiana di Ematologia" (SIE) and of the "European Society for Medical Oncology" (ESMO) The accurate definition of the truly localised forms represents a crucial issue in order to ensure an appropriate treatment design for such patients. The characteristic t(14;18) translocation, which leads to the over-expression of the Bcl-2 gene, is found in approximately 85% of FL; cells bearing this translocation can be detected in the peripheral blood (PB) or bone marrow (BM) by polymerase chain reaction (PCR).

PCR for the t(14;18) translocation provides a sensitive device to identify the presence of minimal non-Hodgkin lymphoma (NHL) cell contamination. Previous experiences have demonstrated that despite the limited stage, Bcl-2/IgH+ cells can be found at diagnosis in PB and/or BM of the majority of the patients. After treatment with local radiotherapy confined to the involved lymph node(s) only, disappearance of circulating Bcl-2/IgH+ cells in PB and/or BM was demonstrated in approximately 60% of positive patients. Quantitative PCR demonstrated the feasibility of clearing PB and BM Bcl-2+ cells after local irradiation of the primary site of the disease only when the basal number of lymphoma cells was <1:100 000.

Anti-CD20 monoclonal antibody treatment has clearly demonstrated, both alone and in combination with chemotherapy and radiotherapy, a high therapeutic potential in FL. A significant impact of treatment with the anti CD20 monoclonal antibody in reducing the minimal residual disease in FL has been demonstrated in several studies when used as consolidation or during the maintenance phase.

No data are currently available concerning the ability of anti-CD20 antibody treatment in reducing the proportion of Bcl-2 positive residual cells after radiotherapy in localized FL. The objective of this study is to take advantage of the therapeutic potential of anti-CD20 monoclonal antibody to reduce or eliminate minimal residual disease in patients with FL in localized stage (I/II) after conventional treatment with local radiotherapy of the involved site(s). The effectiveness of anti-CD20 monoclonal antibody treatment will be determined by the proportion of negativization of residual Bcl-2 positive cells after radiotherapy, evaluated by qualitative and quantitative PCR detection of viable Bcl-2/IgH rearranged cells in PB and/or BM.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed follicular lymphoma grade I-IIIa;
* Stage IA or IIA (no more than 2 contiguous nodal regions) non bulky (<7 cm);
* FLIPI ≤2, FLIPI2 ≤2;
* Previously untreated;
* Age ≥ 18;
* Informed consent;
* Staging with PET-CT, bone marrow biopsy;
* Qualitative/quantitative PCR basal evaluation of Bcl-2/IgH rearranged cells in peripheral blood and bone marrow.

Exclusion Criteria:

* Follicular lymphoma grade IIIb;
* Stage greater than II with more than 2 nodal sites and/or B symptoms and/or bulky disease (>7 cm);
* FLIPI >2, FLIPI2 >2;
* Age < 18;
* Previous treatments for non-Hodgkin's lymphoma;
* Dementia;
* Impossibility to subscribe the informed consent;
* Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones or stable chronic liver disease per investigator assessment);
* Treatment with any known non-marketed drug substance or experimental therapy within 5 terminal half lives or 4 weeks prior to enrollment, whichever is longer, or currently participating in any other interventional clinical study;
* Other past or current malignancy. Subjects who have been free of malignancy for at least 5 years, or have a history of completely resected non-melanoma skin cancer, or successfully treated in situ carcinoma are eligible;
* Chronic or current infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis and active Hepatitis C;
* History of significant cerebrovascular disease in the past 6 months or ongoing event with active symptoms or sequelae;
* Known HIV positive;
* Clinically significant cardiac disease including unstable angina, acute myocardial infarction within six months prior to start of treatment, congestive heart failure (NYHA III-IV), and arrhythmia unless controlled by therapy, with the exception of extra systoles or minor conduction abnormalities;
* Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease which in the opinion of the investigator may represent a risk for the patient;
* Positive serology for Hepatitis B (HB) defined as a positive test for HBsAg. In addition, if negative for HBsAg but HBcAb positive (regardless of HBsAb status), a quantitative HBV-DNA test will be performed and if positive the subject will be excluded. Patients with HBcAb positivity and negative HBV DNA should be prophilactically treated with oral Lamivudine (100 mg /day) in case of treatment with Ofatumumab, to be prosecuted 12 months after treatment;
* Positive serology for hepatitis C (HC) defined as a positive test for HCAb, in which case reflexively perform a HCV-RNA on the same sample to confirm the result;
* Hematologic and blood chemistry exclusion criteria:

  * platelets <50 x 109/L;
  * neutrophils <1.0 x 109/L;
  * creatinine >2.0 times upper normal limit;
  * total bilirubin >1.5 times upper normal limit;
  * ALT >2.5 times upper normal limit;
  * alkaline phosphatase >2.5 times upper normal limit;
* Pregnant or lactating women. Women of childbearing potential must have a negative pregnancy test at screening:

  - Women of childbearing potential, including women whose last menstrual period was less than one year prior to screening, unable or unwilling to use adequate contraception from study start to one year after the last dose of protocol therapy. Adequate contraception is defined as hormonal birth control, intrauterine device, double barrier method or total abstinence;
* Male subjects unable or unwilling to use adequate contraception methods from study start to one year after the last dose of protocol therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-10; Primary Completion 2018-04 (Actual); Study Completion 2022-04-07 (Actual)

PRIMARY OUTCOMES:
Bcl-2 negativization after Ofatumumab | 4 YEARS FROM ENROLLMENT
  The proportion of Bcl-2 negativization after Ofatumumab treatment will be estimated by the proportion, and its confidence interval, of residual Bcl-2 positive cases after radiotherapy, which will became negative after Ofatumumab treatment

SECONDARY OUTCOMES:
Clinical response rate | 4 YEARS FROM ENROLLMENT
  Clinical response rate will be evaluated by the proportion and its confidence interval of patients achieving overall response (OR) complete response (CR) and partial response (PR).
Overall response | 4 YEARS FROM ENROLLMENT
  overall response (OR)
Partial response | 4 YEARS FROM ENROLLMENT
  partial response (PR)
Complete response | 4 YEARS FROM ENROLLMENT
  complete response (CR)
Progression Free Survival | 4 YEARS FROM ENROLLMENT
  Progression Free Survival (PFS) is defined as the length of time between the date of registration and the earliest date of disease progression or death due to any cause; If the patients doesn't not have a documented date of progression or death, the PFS will be censored at the date of last adequate assessment. Relapse Free Survival (RFS) is defined as the length of time between the achievement of Complete Remission (CR) and Relapse of disease
Relapse Free Survival | 4 YEARS FROM ENROLLMENT
  Relapse Free Survival (RFS) is defined as the length of time between the achievement of Complete Remission (CR) and Relapse of disease

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Pulsoni, MD, Study Chair — Policlinico Umberto I - Università "La Sapienza" - Istituto Ematologia
Locations (27):
- Italy (27):
  - Ospedale SS. Antonio e Biagio e Cesare Arrigo, Alessandria, AL
  - Ematologia Azienda Ospedaliera Policlinico, Bari, BA
  - A.O. Spedali Civili, Brescia, BS
  - A.O. Niguarda, Milan, MI
  - Azienda Ospedaliera S. Gerardo Di Monza, Monza, Monza Brianza
  - Osp. S. Maria delle Croci, Ravenna, RA
  - A.O. Bianchi - Melacrino - Morelli, Reggio Calabria, RC
  - Polo Pontino, Latina, Roma
  - Ospedale di Matera, Matera
  - Area Vasta Romagna e IRST, Meldola (FC)
  - Ospedali Riuniti Papardo, Messina
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano, Milan
  - Ospedale S. Raffaele, Milan
  - S.C.D.U Ematologia Azienda Ospedaliero Universitaria Maggiore, Novara
  - U.O. Complessa di Ematologia Ospedale di Parma, Parma
  - IRCCS Policlinico S. Matteo di Pavia, Pavia
  - Ausl Di Piacenza, Piacenza
  - Azienda Ospedaliero Universitaria Pisana U.O. Ematologia, Pisa
  - AO Santa Maria Nuova, Reggio Emilia
  - Ausl Di Rimini, Rimini
  - Ematologia e Trapianto Istituto Regina Elena IFO, Roma
  - Policlinico Umberto I - Università "La Sapienza" - Istituto Ematologia -Dipartimento di Biotecnologie Cellulari ed Ematologia, Roma
  - Ospedale civile DH oncologico, Sassuolo (MO)
  - Policlinico Le Scotte Clinica Ematologica, Siena
  - SC Oncoematologia con autotrapianto AO Santa Maria, Terni
  - A.O. Universitaria Citta' Della Salute E Della Scienza Di Torino, Torino
  - A.O.U. Citta della Salute e della Scienza di Torino, Torino

IPD SHARING:
Plan to Share IPD: Yes
Final study report

REFERENCES:
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Abbott BL. Chronic lymphocytic leukemia: recent advances in diagnosis and treatment. Oncologist. 2006 Jan;11(1):21-30. doi: 10.1634/theoncologist.11-1-21. PMID 16401710
- [Background] Apostolidis J, Gupta RK, Grenzelias D, Johnson PW, Pappa VI, Summers KE, Salam A, Adams K, Norton AJ, Amess JA, Matthews J, Bradburn M, Lister TA, Rohatiner AZ. High-dose therapy with autologous bone marrow support as consolidation of remission in follicular lymphoma: long-term clinical and molecular follow-up. J Clin Oncol. 2000 Feb;18(3):527-36. doi: 10.1200/JCO.2000.18.3.527. PMID 10653868
- [Background] Armitage JO, Weisenburger DD. New approach to classifying non-Hodgkin's lymphomas: clinical features of the major histologic subtypes. Non-Hodgkin's Lymphoma Classification Project. J Clin Oncol. 1998 Aug;16(8):2780-95. doi: 10.1200/JCO.1998.16.8.2780. PMID 9704731
- [Background] Barosi G, Carella A, Lazzarino M, Marchetti M, Martelli M, Rambaldi A, Tarella C, Vitolo U, Zinzani PL, Tura S. Management of nodal indolent (non marginal-zone) non-Hodgkin's lymphomas: practice guidelines from the Italian Society of Hematology, Italian Society of Experimental Hematology and Italian Group for Bone Marrow Transplantation. Haematologica. 2005 Sep;90(9):1236-57. PMID 16154848
- [Background] Berinstein NL, Reis MD, Ngan BY, Sawka CA, Jamal HH, Kuzniar B. Detection of occult lymphoma in the peripheral blood and bone marrow of patients with untreated early-stage and advanced-stage follicular lymphoma. J Clin Oncol. 1993 Jul;11(7):1344-52. doi: 10.1200/JCO.1993.11.7.1344. PMID 8315432
- [Background] Binet JL, Caligaris-Cappio F, Catovsky D, Cheson B, Davis T, Dighiero G, Dohner H, Hallek M, Hillmen P, Keating M, Montserrat E, Kipps TJ, Rai K; International Workshop on Chronic Lymphocytic Leukemia (IWCLL). Perspectives on the use of new diagnostic tools in the treatment of chronic lymphocytic leukemia. Blood. 2006 Feb 1;107(3):859-61. doi: 10.1182/blood-2005-04-1677. Epub 2005 Oct 13. PMID 16223776
- [Background] Binet JL, Auquier A, Dighiero G, Chastang C, Piguet H, Goasguen J, Vaugier G, Potron G, Colona P, Oberling F, Thomas M, Tchernia G, Jacquillat C, Boivin P, Lesty C, Duault MT, Monconduit M, Belabbes S, Gremy F. A new prognostic classification of chronic lymphocytic leukemia derived from a multivariate survival analysis. Cancer. 1981 Jul 1;48(1):198-206. doi: 10.1002/1097-0142(19810701)48:13.0.co;2-v. PMID 7237385
- [Background] Weiss LM, Warnke RA, Sklar J, Cleary ML. Molecular analysis of the t(14;18) chromosomal translocation in malignant lymphomas. N Engl J Med. 1987 Nov 5;317(19):1185-9. doi: 10.1056/NEJM198711053171904. PMID 3657890
- [Background] Brown JR, Feng Y, Gribben JG, Neuberg D, Fisher DC, Mauch P, Nadler LM, Freedman AS. Long-term survival after autologous bone marrow transplantation for follicular lymphoma in first remission. Biol Blood Marrow Transplant. 2007 Sep;13(9):1057-65. doi: 10.1016/j.bbmt.2007.05.012. Epub 2007 Jul 16. PMID 17697968
- [Background] Ygge J. [Acute heparin therapy--standard dose or dosage according to individual sensitivity?]. Lakartidningen. 1977 Mar 9;74(10):921-4. No abstract available. Swedish. PMID 839876
- [Background] Gribben JG, Freedman AS, Neuberg D, Roy DC, Blake KW, Woo SD, Grossbard ML, Rabinowe SN, Coral F, Freeman GJ, et al. Immunologic purging of marrow assessed by PCR before autologous bone marrow transplantation for B-cell lymphoma. N Engl J Med. 1991 Nov 28;325(22):1525-33. doi: 10.1056/NEJM199111283252201. PMID 1944436
- [Background] Chao DT, Korsmeyer SJ. BCL-2 family: regulators of cell death. Annu Rev Immunol. 1998;16:395-419. doi: 10.1146/annurev.immunol.16.1.395. PMID 9597135
- [Background] Corradini P, Ladetto M, Zallio F, Astolfi M, Rizzo E, Sametti S, Cuttica A, Rosato R, Farina L, Boccadoro M, Benedetti F, Pileri A, Tarella C. Long-term follow-up of indolent lymphoma patients treated with high-dose sequential chemotherapy and autografting: evidence that durable molecular and clinical remission frequently can be attained only in follicular subtypes. J Clin Oncol. 2004 Apr 15;22(8):1460-8. doi: 10.1200/JCO.2004.10.054. PMID 15084619
- [Background] Lopez-Guillermo A, Cabanillas F, McDonnell TI, McLaughlin P, Smith T, Pugh W, Hagemeister F, Rodriguez MA, Romaguera JE, Younes A, Sarris AH, Preti HA, Lee MS. Correlation of bcl-2 rearrangement with clinical characteristics and outcome in indolent follicular lymphoma. Blood. 1999 May 1;93(9):3081-7. PMID 10216105
- [Background] Rambaldi A, Lazzari M, Manzoni C, Carlotti E, Arcaini L, Baccarani M, Barbui T, Bernasconi C, Dastoli G, Fuga G, Gamba E, Gargantini L, Gattei V, Lauria F, Lazzarino M, Mandelli F, Morra E, Pulsoni A, Ribersani M, Rossi-Ferrini PL, Rupolo M, Tura S, Zagonel V, Zaja F, Zinzani P, Reato G, Foa R. Monitoring of minimal residual disease after CHOP and rituximab in previously untreated patients with follicular lymphoma. Blood. 2002 Feb 1;99(3):856-62. doi: 10.1182/blood.v99.3.856. PMID 11806987
- [Background] van Oers MH, Klasa R, Marcus RE, Wolf M, Kimby E, Gascoyne RD, Jack A, Van't Veer M, Vranovsky A, Holte H, van Glabbeke M, Teodorovic I, Rozewicz C, Hagenbeek A. Rituximab maintenance improves clinical outcome of relapsed/resistant follicular non-Hodgkin lymphoma in patients both with and without rituximab during induction: results of a prospective randomized phase 3 intergroup trial. Blood. 2006 Nov 15;108(10):3295-301. doi: 10.1182/blood-2006-05-021113. Epub 2006 Jul 27. PMID 16873669
- [Background] Pulsoni A, Starza ID, Frattarelli N, Ghia E, Carlotti E, Cavalieri E, Matturro A, Tempera S, Rambaldi A, Foa R. Stage I/II follicular lymphoma: spread of bcl-2/IgH+ cells in blood and bone marrow from primary site of disease and possibility of clearance after involved field radiotherapy. Br J Haematol. 2007 May;137(3):216-20. doi: 10.1111/j.1365-2141.2007.06545.x. PMID 17408460